CLINICAL TRIAL: NCT02786121
Title: Is Kinesiophobia a Predictive Factor of the Early Functional Recovery After Total Hip Replacement? - An Observational Study
Brief Title: The Role of Kinesiophobia in the Functional Recovery After Hip Replacement
Acronym: kinesiofob
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0008317
Record Dates: First submitted 2016-04-15; First posted 2016-05-30 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Hip Osteoarthritis
Keywords: hip replacement,; rehabilitation,; early ambulation,
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Several authors explain as the kinesiophobia plays an important role for the recovery after orthopaedic surgery. The aim of the investigators study is to investigate if the kinesiophobia is able to influence the early recovery after total hip arthroplasty. The early recovery will be measured by the ILOA Score. The Tampa Scale of Kinesiophobia will measure the fear level of movement. All the other variable that could influence the ILOA Score are identified and collected: age, sex, body max index, ability of patient pre-surgery, type of anesthesia, length of stay, pain, haemoglobin, possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip joint replacement
* Clinical symptoms from more than 3 months

Exclusion Criteria:

* other orthopaedic surgery on the lower limb In the last year
* Not italian speaking
* Hip arthroplasty following fractures, revision surgery, and partial replacement
* Patients with concomitant neurologic (Parkinson, ictus), rheumatologic (rheumatoid arthritis) diseases,
* cognitive impaired.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total hip arthroplasties patients following chronic joint disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Iowa Level of Assistance (ILOA) Score | 5 days after surgery
  The outcome considered was the level of autonomy achieved by the patients at the 5th days after surgery, measured by the Iowa Level of Assistance (ILOA) scale that took into account the patient's autonomy in carrying out functional 5 activities: supine-to-sitting, sitting-to-standing, walking, climbing 3 steps, and gait speed. The total score ranged from 0 to 50, where 0 was the patient's complete autonomy and 50 the maximum dependence. The score was based on the level of help that was supplied to the patient by the operator for the safe execution of activities, with a range between 0 and 30, and the type of assistive device used with a range between 0 and 20. The physiotherapist will collect the ILOA Score.

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Morri, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morri M, Venturini E, Franchini N, Ruisi R, Culcasi A, Ruggiero A, Govoni C, Benedetti MG. Is kinesiophobia a predictor of early functional performance after total hip replacement? A prospective prognostic cohort study. BMC Musculoskelet Disord. 2020 Nov 7;21(1):724. doi: 10.1186/s12891-020-03748-7. PMID 33160343